CLINICAL TRIAL: NCT00937313
Title: The Pharmacokinetics and Potential Health Effects of Champagne Wine in Human Subjects
Status: Completed | Type: Observational
Sponsor: University of Reading (Other)
Responsible Party: Jeremy Paul Edward Spencer, PhD, Department of Food and Nutritional Sciences
Other Study IDs: UoR 07/16
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: No Condition. Assessment of Healthy Volunteers.

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — plasma serum urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Champagne wine
  Interventions: Other: Champagne wine intervention
- Placebo: alcohol with sparkling mineral water
  Interventions: Other: Champagne wine intervention

INTERVENTIONS:
Other: Champagne wine intervention — Placebo-controlled randomised cross-over human trial
  Other Names: Non applicable

SUMMARY:
* To assess whether acute, moderate Champagne wine consumption modulates endothelial function in healthy human volunteers.
* To establish the bioavailability of Champagne wine polyphenols and their metabolism.

DETAILED DESCRIPTION:
Subjects refrained from consuming high polyphenol foods for 48 h prior to the start of the study and for 32 h post initiation. In particular, the following foods and beverages were excluded from volunteer diets: cocoa containing products, coffee, tea and wine. The study was designed as a single blind, randomized, crossover intervention trial, where volunteers were asked to consume either 375 ml of Champagne wine or a placebo matched for alcohol content, sugars and fruit-derived acids. Subjects were assessed for anthropometric measurements and provided a urine sample prior baseline Laser Doppler Imaging with iontophoresis (LDI) measurements. Subjects were then cannulated and a baseline blood sample was collected. Subjects were then randomly assigned to either the Champagne wine or placebo group and asked to consume the beverage within a 10 min period. Following a standardised breakfast blood samples were collected at: 15, 30, 45, 60, 120, 180, 240, 300, 360 and 480 minutes post consumption and pooled urine samples were collected over 3 x 8 h periods. A standardised breakfast and lunch were also consumed at 15 and 200 minutes post beverage. LDI measurements were carried out at 120, 240, 360 and 480 minutes. Subjects also provided 24 h and 32 h blood and urine samples. Following a washout period of 28 days, volunteers returned to the unit to complete the second arm of the study where the procedure above was repeated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, aged between 20 and 65 years, with a Body Mass Index (BMI) between 19 and 25 kg/m². Normal concentrations of liver enzymes (AST, ALT, gamma GT), normal hemoglobin, hematocrit and leucocyte counts and an absence of glucose and protein in urine

Exclusion Criteria:

* Individuals with diabetes, any form of liver or gastrointestinal disorder, low BMI (<19), high blood pressure (>150/90 mm/Hg), anaemia, gall bladder problems, present illness, or those taking dietary supplements, vigorous exercise (> 3 x 20 min/week), or alcohol consumption more than 120 g (women) and 168 g (men) per week , pregnant or lactating females.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2007-07; Primary Completion 2008-02 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Assessment of endothelial function by Laser Doppler Imaging with iontophoresis. Blood Assessment of lipid profile, inflammatory markers, plasma antioxidant and oxidant capacity, liver enzyme and metalloproteinase blood concentrations. | 6 months

SECONDARY OUTCOMES:
Bioavailability of phytochemicals and metabolite excretion. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy PE Spencer, PhD, Principal Investigator — The University of Reading; David Vauzour, PhD, Principal Investigator — The University of Reading; Julie Lovegrove, PhD, Principal Investigator — The University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, Reading, Berkshire, United Kingdom